CLINICAL TRIAL: NCT01789372
Title: Effects of Mediyoga in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Maria Nilsson, Reg nurse, Danderyd Hospital
Other Study IDs: YOGAFF-001
Record Dates: First submitted 2013-02-05; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; yoga; quality of life; blood pressure; heart rate; heart rate variability
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determinate if mediyoga has effects in quality of life, heart rate variability, blood pressure , heart rate in patients with paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
This is randomized prospective pilot study. Eighty patients from Danderyd hospital, Stockholm, Sweden were randomized to either mediyoga group or control group. The mediyoga group were completing yoga for one hour, once a week for 12 weeks together with usual treatment. The controlgroup had only usual treatment.The usual treatment consists of pharmaceutical, cardio version and ablation. Quality of life ( SF-36, EQ-5d), blood pressure, heart rate and 24-hours ekokardiografi were measured at baseline and after twelve weeks.A follow up after six months was accomplished with SF-36 and EQ-5d, bloodpressure and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAF

Exclusion Criteria:

* The exclusions criteria were multiple concurrent medical conditions and/or cognitive dysfunction (in the diagnosis of e.g. mental illness), considered not to be able to carry out yoga owing to ability to move and those who have difficulties to understand the Swedish language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic. All participants should have been on usual treatment (medication, cardio version or ablation) for at least three months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | Change from baseline in SF-36 after 12 weeks.Change from baseline in SF-36 after six months.
Quality of life | Change from baseline in SF-36 after 12 weeks.Change from baseline in EQ-5D after six month

SECONDARY OUTCOMES:
Blood pressure | Change from baseline in blood pressure after 12 weeks. Change from baseline in blood pressure after six months
heart rate | Change from baseline in heart rate after 12 weeks.Change from baseline in heart rate after six months.
Heart variability | Change from baseline in heart variability after 12 weeks.Change from baseline in heart variability after six months.

CONTACTS AND LOCATIONS:
Overall Officials: Viveka Frykman, Phd, MD, Study Director — Danderyd hospital, Karolinska Institute Sweden
Locations (1):
- Danderyds hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Wahlstrom M, Medin J, Karlsson MR. Gender differences in health-related quality of life, blood pressure and heart rate among patients with paroxysmal atrial fibrillation after performing MediYoga. Int J Cardiol Heart Vasc. 2023 Sep 22;49:101274. doi: 10.1016/j.ijcha.2023.101274. eCollection 2023 Dec. PMID 37766884